CLINICAL TRIAL: NCT00080665
Title: A Phase I Study Of Weekly Taxotere (Docetaxel) And Gleevec (STI571, Imatinib Mesylate, CGP 57148B) In Locally Advanced Or Metastatic Breast Cancer
Brief Title: Docetaxel and Imatinib Mesylate in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0214 CDR0000354504; P30CA006973 (NIH); JHOC-J0214 (Other: SKCCC at Johns Hopkins); SKCCC-J0214 (Other: SKCCC at Johns Hopkins)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: male breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Docetaxel; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib mesylate and docetaxel (Experimental): Imatinib mesylate (400-600 mg, oral, once daily) and docetaxel (15-30 mg/m2, IV, weekly on days 1, 8, and 15) each 28 day cycle
  Interventions: Drug: docetaxel; Drug: imatinib mesylate

INTERVENTIONS:
Drug: docetaxel — Docetaxel (15-30 mg/m2, IV, weekly on days 1, 8, and 15) each 28 day cycle
  Other Names: Taxotere
Drug: imatinib mesylate — Imatinib mesylate (400-600 mg, oral, once daily) each 28 day cycle
  Other Names: Gleevec, STI571

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as docetaxel work in different ways to stop tumor cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving docetaxel with imatinib mesylate may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel when given together with imatinib mesylate in treating patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety profile, maximum tolerated dose, and recommended phase II dose of docetaxel when administered with imatinib mesylate in patients with locally advanced or metastatic breast cancer.

Secondary

* Determine the pharmacokinetic profile of this regimen in these patients.
* Determine the potential effects of this regimen on CYP3A4 activity and docetaxel metabolism in these patients.
* Correlate docetaxel and imatinib mesylate exposure (utilizing total and unbound docetaxel and imatinib mesylate plasma concentrations) with drug response (e.g., pharmacodynamic effects, drug toxicity, and response) in these patients.
* Determine response rate, duration of response, and time to treatment failure in patients treated with this regimen.
* Correlate proteomic profile changes in serum with tumor burden and response in patients treated with this regimen.
* Correlate pharmacokinetic parameters, tissue expression of specific receptor tyrosine kinases (e.g., c-Kit, platelet-derived growth factor receptor [PDGFR], and phosphorylated PDGFR) in paraffin blocks, and pharmacodynamic assays with antitumor activity of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of docetaxel.

Patients receive docetaxel IV over 1 hour on days 1, 8, and 15 and oral imatinib mesylate (STI571) on days 8-28 of course 1 and days 1-28 of all subsequent courses. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity*. Patients with stable or responding disease after at least 2 courses of therapy may discontinue docetaxel and continue therapy with single-agent STI571 until disease progression.

NOTE: *Patients experiencing excessive docetaxel-related toxicity who have completed at least 2 full courses may continue on single-agent STI571 in the absence of disease progression or excessive STI571-related toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional cohort of 6-12 patients receives treatment at the MTD.

Patients are followed at 30 days.

PROJECTED ACCRUAL: Approximately of 18-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Stage IIIB, IIIC, or IV disease
* Measurable or evaluable disease
* Stable brain metastases allowed provided prior surgery or radiotherapy was completed more than 90 days ago
* No documented or suspected leptomeningeal disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ upper limit of normal (ULN)
* Meets 1 of the following criteria for AST or ALT AND alkaline phosphatase:

  * AST or ALT ≤ ULN AND alkaline phosphatase ≤ 5 times ULN
  * AST or ALT ≤ 2.5 times ULN AND alkaline phosphatase ≤ ULN
  * AST or ALT ≤ 1.5 times ULN AND alkaline phosphatase ≤ 2.5 times ULN
* No known acute or chronic liver disease (e.g., chronic active hepatitis or cirrhosis)

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No New York Heart Association class III or IV heart disease
* No congestive heart failure
* No myocardial infarction within the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation
* No other primary malignancy except those malignancies that are clinically insignificant AND do not require active intervention
* No other concurrent severe and/or life-threatening medical disease
* No significant history of noncompliance to medical regimens or inability to grant reliable informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 14 days since prior systemic trastuzumab (Herceptin®)
* No concurrent trastuzumab
* No concurrent biologic therapy for the primary malignancy

Chemotherapy

* Prior taxane therapy, including docetaxel, in the adjuvant or metastatic setting allowed
* At least 21 days since prior systemic chemotherapy (14 days for weekly or oral chemotherapy and 42 days for nitrosoureas or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy

* At least 14 days since prior systemic hormonal therapy
* No concurrent antiestrogen therapy
* No concurrent routine systemic corticosteroid therapy except as premedication for chemotherapy
* Concurrent megestrol allowed only as an appetite stimulant

Radiotherapy

* See Disease Characteristics
* At least 14 days since prior radiotherapy
* No prior radiotherapy to only site of measurable/evaluable disease unless there is new evidence of post-radiotherapy disease progression
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* More than 2 weeks since prior major surgery

Other

* Recovered from all prior therapy
* At least 14 days since prior daily or weekly systemic investigational treatment
* No concurrent warfarin for full anticoagulation

  * Concurrent low-dose warfarin (e.g., 1 mg/day) allowed for prophylaxis of central venous access
* No concurrent treatment with any of the following:

  * Phenobarbital
  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Hypericum perforatum (St. John's wort)
* No other concurrent therapies for the primary malignancy
* No other concurrent investigational drugs or systemic therapy
* No concurrent bisphosphonates unless started before study therapy
* No concurrent grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-12; Primary Completion 2007-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
2.1.1 To determine the safety profile, maximum tolerated dose, and recommended dose for subsequent phase II studies of a combination regimen of daily STI571 with weekly docetaxel on days 1, 8, and 15 in a 28-day cycle. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. Wolff, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Connolly RM, Rudek MA, Garrett-Mayer E, Jeter SC, Donehower MG, Wright LA, Zhao M, Fetting JH, Emens LA, Stearns V, Davidson NE, Baker SD, Wolff AC. Docetaxel metabolism is not altered by imatinib: findings from an early phase study in metastatic breast cancer. Breast Cancer Res Treat. 2011 May;127(1):153-62. doi: 10.1007/s10549-011-1413-6. Epub 2011 Feb 25. PMID 21350820
- [Derived] Fackler MJ, Lopez Bujanda Z, Umbricht C, Teo WW, Cho S, Zhang Z, Visvanathan K, Jeter S, Argani P, Wang C, Lyman JP, de Brot M, Ingle JN, Boughey J, McGuire K, King TA, Carey LA, Cope L, Wolff AC, Sukumar S. Novel methylated biomarkers and a robust assay to detect circulating tumor DNA in metastatic breast cancer. Cancer Res. 2014 Apr 15;74(8):2160-70. doi: 10.1158/0008-5472.CAN-13-3392. PMID 24737128